CLINICAL TRIAL: NCT02139228
Title: A Phase IIIb, Controlled, Open Label, Single-Center, Persistency, Extension Study in Chinese Children After a 2+1 Dose Series of Either CRM197-Conjugate Haemophilus Influenzae Type b Vaccine or Tetanus Toxoid-Conjugate Haemophilus Influenzae Type b Vaccine
Brief Title: Persistency Study After Hib-CRM (Cross-Reacting Material)197 or Hib-TT (Tetanus Toxoid) Vaccines in Chinese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V37_07E2
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-10

CONDITIONS: Meningitis, Epiglottitis, Pneumonia, Arthritis Caused by Haemophilus Influenzae Type b
Keywords: Haemophilus influenzae type b; persistency; children; CRM197; anti-PRP antibody
MeSH Terms: conditions — Meningitis; Epiglottitis; Pneumonia; Haemophilus Infections | interventions — HibTITER protein, Haemophilus influenzae; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hib CRM197 (Experimental): Subjects treated with 3 doses of CRM 197 -conjugate Haemophilus influenzae type b vaccine (study vaccine): 2 doses given one month apart during study V37_07 (NCT01044316) and a booster dose of the same vaccine six months after, during study V37_07E1 (NCT01226953).
  No vaccine was administered during this trial
  Interventions: Biological: Hib-CRM197
- Hib TT (Active Comparator): Subjects treated with 3 doses of Tetanus Toxoid-conjugate Haemophilus influenzae type b vaccine (comparator vaccine): 2 doses given one month apart during study V37_07 (NCT01044316) and a booster dose of the same vaccine six months after, during study V37_07E1 (NCT01226953).
  No vaccine was administered during this trial
  Interventions: Biological: Hib-TT

INTERVENTIONS:
Biological: Hib-CRM197 — No vaccine administered in V37_07E2 study
  Arms: Hib CRM197
Biological: Hib-TT — No vaccine administered in V37_07E2 study
  Arms: Hib TT

SUMMARY:
Evaluate the persistency of immune response against Haemophilus influenzae type b by assessing anti-PRP antibody levels in children vaccinated with either Hib-CRM197 or Hib-TT booster vaccine approximately 4 years before.

ELIGIBILITY:
Inclusion Criteria:

1. Children previously enrolled in V37_07E1 study and who received the appropriate vaccination.
2. Children whose parent(s) or legal guardian(s) had given written consent after the nature of the study was explained according to local regulatory requirements.

Exclusion Criteria:

1. Any confirmed or suspected current immunosuppressive or immunodeficient condition since the end of V37_07E1 study, based on medical history and physical examination (no laboratory testing required).
2. Treatment with corticosteroids or other immunosuppressive/immunostimulant drugs as defined below:

   i) chronic use of oral and parenteral immunosuppressants (>= 15 days of use) or other immune-modifying drugs within 60 days prior to the blood sampling (short term usage of topical, inhaled and/or intranasal corticosteroids were allowed) ii) receipt of immunostimulants within 60 days prior to Visit 1
3. Administration of immunoglobulins and/or any blood products up to 3 months before enrollment.
4. Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the blood sampling.
5. Any condition, which, in the opinion of the investigator, might be a contraindication to the execution of the blood draw.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 426 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- DingXing Center for Disease Control and Prevention, Dingxing, Hebei, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One center in China
Pre-assignment Details: All subjects enrolled into the parent V37_07E1 study were invited to participate in the trial.
Period: Overall Study
Arm/Group | Hib CRM197 | Hib TT
Started | 215 | 211
Completed | 215 | 211
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hib CRM197 | Hib TT | Total
Number analyzed (Participants) | 215 | 211 | 426
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 5 (0) | 5 (0) | 5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 106 | 205
  Male | 116 | 105 | 221

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Anti-PRP (Polyribosyl Ribitol Phosphate) Concentrations at Day 1 (4 Years Post Booster Dose Administered in Study V37_07E1)
Description: Immunogenicity was measured as geometric mean of Anti- PRP Concentrations, approximately 4 years after booster vaccination with either Hib-CRM197 or Hib-TT in children participating in previous V37_07E1 trial.
Time Frame: At Day 1 (4 years post booster dose administered in study V37_07E1)
Population: Analysis was evaluated on the Per Protocol set (PPS)-All subjects in the All Enrolled Set with no reportable protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: Concentration in μg/mL
Arm/Group | Hib CRM197 | Hib TT
Number analyzed (Participants) | 215 | 211
Concentration in μg/mL | 2.66 [2 to 3.54] | 5.05 [3.97 to 6.42]
Statistical Analysis 1: Comparison: Hib CRM197 vs Hib TT; Test type: Superiority or Other; ANOVA; Vaccine Group Ratios = 0.53, 95% CI 2-sided [0.36 to 0.76]

2. Secondary Outcome: Percentages of Subjects With Anti-PRP Concentrations ≥1.0 μg/mL and ≥0.15 μg/mL at Day 1 (4 Years Post Booster Dose Administered in Study V37_07E1)
Description: Immunogenicity was measured as the percentages of subjects with Anti-PRP Concentrations ≥1.0 μg/mL and ≥0.15 μg/mL approximately 4 years after booster vaccination with either Hib-CRM197 or Hib-TT in V37_07E1 trial.
Time Frame: At Day 1 (4 years post booster dose administered in study V37_07E1)
Population: Analysis was evaluated on the Per Protocol set (PPS) (i.e. All subjects in the All Enrolled Set with no reportable protocol deviations).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Hib CRM197 | Hib TT
Number analyzed (Participants) | 215 | 211
Percentage of subjects
  Anti-PRP Concentrations ≥ 1.0 μg/mL | 77 [71 to 82] | 88 [83 to 92]
  Anti-PRP Concentrations ≥ 0.15 μg/mL | 77 [71 to 82] | 88 [83 to 92]
Statistical Analysis 1: Comparison: Hib CRM197 vs Hib TT; Test type: Superiority or Other; Clopper-Pearson; Vaccine Group Differences = -11, 95% CI 2-sided [-18.6 to -4.2]

ADVERSE EVENTS:
Description: Safety section not applicable for this study
Arm/Group | Hib CRM197 | Hib TT
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement: The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.